CLINICAL TRIAL: NCT01239797
Title: Phase 3, Randomized, Open Label Trial of Lenalidomide/Dexamethasone With or Without Elotuzumab in Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: Phase III Study of Lenalidomide and Dexamethasone With or Without Elotuzumab to Treat Relapsed or Refractory Multiple Myeloma
Acronym: ELOQUENT - 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-004; 2010-020347-12 (EudraCT Number)
Record Dates: First submitted 2010-11-08; First posted 2010-11-11 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenalidomide + Dexamethasone (Active Comparator)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- Lenalidomide + Dexamethasone +Elotuzumab (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone (Oral); Drug: Dexamethasone (IV); Biological: Elotuzumab (BMS-901608; HuLuc63)

INTERVENTIONS:
Drug: Lenalidomide — Capsules, Oral, 25 mg, once daily, on Days 1-21, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Revlimid®
Drug: Dexamethasone — Tablets, Oral, 40 mg, weekly, on Days 1, 8, 15, 22, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone
Drug: Dexamethasone (Oral) — On weeks without Elotuzumab dosing: Tablets, Oral, 40mg, Repeat every 28 days until subject meets criteria for discontinuation of study drug.
  On weeks with Elotuzumab dosing: Tablets, Oral, 28 mg, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone +Elotuzumab
Drug: Dexamethasone (IV) — On weeks without Elotuzumab dosing: Not Applicable (N/A)
  On weeks with Elotuzumab dosing: Solution, Intravenous (IV), 8 mg, weekly, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone +Elotuzumab
Biological: Elotuzumab (BMS-901608; HuLuc63) — Solution, IV, 10 mg/kg, weekly, on Days 1, 8, 15, 22 (cycles 1&2); Days 1 and 15 (cycles 3 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Arms: Lenalidomide + Dexamethasone +Elotuzumab

SUMMARY:
The purpose of the study is to determine whether the addition of Elotuzumab to Lenalidomide/low-dose Dexamethasone will increase the progression free survival (PFS).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Documented progression from most recent line of therapy
* 1-3 prior lines of therapy
* Measurable disease
* Life expectancy ≥3 months
* Prior treatment with Lenalidomide permitted if:

  1. Best response achieved was ≥Partial Response (PR)
  2. Patient was not refractory
  3. Patient did not discontinue due to a Grade ≥3 related adverse event
  4. Subject did not receive more than 9 cycles of Lenalidomide and had at least 9 months between the last dose of Lenalidomide and progression

Exclusion Criteria:

* Subjects with non-secretory or oligo-secretory or serum free light-chain only myeloma
* Active plasma cell leukemia
* Known Human immunodeficiency virus (HIV) infection or active hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2014-09-02 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (202):
- United States (62):
  - Northwest Alabama Cancer Center, Pc, Muscle Shoals, Alabama
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Local Institution, Berkeley, California
  - Local Institution, Burbank, California
  - Compassionate Cancer Res Grp, Corona, California
  - Local Institution, Corona, California
  - San Diego Pacific Oncology& Hematology Associates, Inc, Encinitas, California
  - Local Institution, Greenbrae, California
  - Ucla-Division Of Hematology/Oncology, Los Angeles, California
  - Medical Oncology Care Associates, Orange, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Local Institution, Vallejo, California
  - Local Institution, Boca Raton, Florida
  - Cancer Care Centers Of Florida, Brooksville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Local Institution, New Port Richey, Florida
  - Cancer Institute Of Florida, Orlando, Florida
  - Local Institution, Titusville, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - Georgia Health Science University, Augusta, Georgia
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Mishawaka, Indiana
  - Local Institution, Iowa City, Iowa
  - Local Institution, Lexington, Kentucky
  - Local Institution, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Cancer Center Of Acadiana At Lafayette General, Lafayette, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Dana Farber Cancer Inst, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Capitol Comprehensive Cancer Care Center, Jefferson City, Missouri
  - Local Institution, Springfield, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - NYU Clinical Cancer Center, New York, New York
  - Local Institution, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Local Institution, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Gaston Hematology & Oncology, Gastonia, North Carolina
  - Local Institution, Bismarck, North Dakota
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Bethlehem, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Greenville, South Carolina
  - Local Institution, Knoxville, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists Of South Texas, Pa, Corpus Christi, Texas
  - Ut Southwestern Medical Center, Dallas, Texas
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Hematology-Oncology Associates Of Fredricksburg, Inc, Fredericksburg, Virginia
  - Va Puget Sound Health Care System, Seattle, Washington
  - Gundersen Clinic, Ltd, La Crosse, Wisconsin
  - University Of Wisconsin Hospital And Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Local Institution, Albury, New South Wales
  - Local Institution, Canberra, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Malvern, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Nedlands, Western Australia
  - Local Institution, Murdoch
- Austria (4):
  - Local Institution, Rankweil
  - Local Institution, Steyr
  - Local Institution, Vienna
  - Local Institution, Wels
- Belgium (6):
  - Local Institution, Antwerp
  - Local Institution, Brussels
  - Local Institution, Brussles
  - Local Institution, Edegem-antwerp
  - Local Institution, Liège
  - Local Institution, Yvoir
- Canada (9):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, London, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
  - Local Institution, Barrie
  - Local Institution, Montreal
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Copenhagen
  - Local Institution, Odense C
  - Local Institution, Vejle
- France (14):
  - Local Institution, Blois
  - Local Institution, Bordeaux
  - Local Institution, Caen
  - Local Institution, Clamart
  - Local Institution, La Roche-sur-Yon
  - Local Institution, La Tronche
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pierre Benita
  - Local Institution, Toulouse
  - Local Institution, Tours
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (17):
  - Local Institution, Aschaffenburg
  - Local Institution, Berlin
  - Local Institution, Chemnitz
  - Local Institution, Cologne
  - Local Institution, Dresden
  - Local Institution, Hamburg
  - Local Institution, Hamm
  - Local Institution, Heidelberg
  - Local Institution, Jena
  - Local Institution, Kiel
  - Local Institution, Marburg
  - Local Institution, München
  - Local Institution, Münster
  - Local Institution, Ravensburg
  - Local Institution, Tübingen
  - Local Institution, Ulm
  - Local Institution, Würzburg
- Greece (3):
  - Local Institution, Athens
  - Local Institution, Ioannina
  - Local Institution, Larissa
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Győr
  - Local Institution, Szeged
- Ireland (2):
  - Local Institution, Dublin
  - Local Institution, Tullamore
- Israel (5):
  - Local Institution, Afula
  - Local Institution, Jerusalem
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Ẕerifin
- Italy (12):
  - Local Institution, Ancona
  - Local Institution, Bergamo
  - Local Institution, Bologna
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Meldola
  - Local Institution, Milan
  - Local Institution, Palermo
  - Local Institution, Ravenna
  - Local Institution, Rimini
  - Local Institution, Roma
  - Local Institution, Torino
- Japan (17):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Maebashi, Gunma
  - Local Institution, Shibukawa-shi, Gunma
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Sendai, Miyagi
  - Local Institution, Osaka, Osaka
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Koto-ku, Tokyo
  - Local Institution, Shibuya-ku, Tokyo
  - Local Institution, Shinjuuku-ku, Tokyo
  - Local Institution, Kamogawa, Toyko
  - Local Institution, Chiba
  - Local Institution, Fukuoka
  - Local Institution, Kyoto
  - Local Institution, Niigata
  - Local Institution, Okayama
  - Local Institution, Toyohashi
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Chorzów
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, San Juan
- Romania (3):
  - Local Institution, Brasov
  - Local Institution, Bucaresti
  - Local Institution, Bucharest
- Spain (6):
  - Local Institution, Badalona-Barcelona
  - Local Institution, Madrid
  - Local Institution, Murcia
  - Local Institution, Salamanca
  - Local Institution, Santiago de Comp-coruna
  - Local Institution, Toledo
- Switzerland (2):
  - Local Institution, Bern
  - Local Institution, Geneva
- Turkey (Türkiye) (4):
  - Local Institution, Izmir, Bornova
  - Local Institution, Istanbul, CAPA
  - Local Institution, Ankara
  - Local Institution, Izmir
- Local Institution, Leicester, United Arab Emirates
- United Kingdom (9):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Airdrie, Lancashire
  - Local Institution, Edinburgh, Midlothian
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Sutton, Surrey
  - Local Institution, Leeds
  - Local Institution, London
  - Local Institution, Newcastle upon Tyne

REFERENCES:
- [Derived] Dimopoulos MA, Lonial S, Betts KA, Chen C, Zichlin ML, Brun A, Signorovitch JE, Makenbaeva D, Mekan S, Sy O, Weisel K, Richardson PG. Elotuzumab plus lenalidomide and dexamethasone in relapsed/refractory multiple myeloma: Extended 4-year follow-up and analysis of relative progression-free survival from the randomized ELOQUENT-2 trial. Cancer. 2018 Oct 15;124(20):4032-4043. doi: 10.1002/cncr.31680. Epub 2018 Sep 11. PMID 30204239
- [Derived] Passey C, Mora J, Dodge R, Gibiansky L, Sheng J, Roy A, Bello A, Gupta M. An Integrated Assessment of the Effects of Immunogenicity on the Pharmacokinetics, Safety, and Efficacy of Elotuzumab. AAPS J. 2017 Mar;19(2):557-567. doi: 10.1208/s12248-016-0033-9. Epub 2017 Jan 9. PMID 28070715
- [Derived] Lonial S, Dimopoulos M, Palumbo A, White D, Grosicki S, Spicka I, Walter-Croneck A, Moreau P, Mateos MV, Magen H, Belch A, Reece D, Beksac M, Spencer A, Oakervee H, Orlowski RZ, Taniwaki M, Rollig C, Einsele H, Wu KL, Singhal A, San-Miguel J, Matsumoto M, Katz J, Bleickardt E, Poulart V, Anderson KC, Richardson P; ELOQUENT-2 Investigators. Elotuzumab Therapy for Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2015 Aug 13;373(7):621-31. doi: 10.1056/NEJMoa1505654. Epub 2015 Jun 2. PMID 26035255
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 646 participants were randomized and 635 were treated
Groups:
- Lenalidomide + Dexamethasone + Elotuzumab: Lenalidomide: Capsules, Oral, 25 mg, once daily, on Days 1-21 Repeat every 28 days until participants met criteria for discontinuation of study drug Dexamethasone (Oral): On weeks without Elotuzumab dosing: Tablets, Oral, 40mg Repeat every 28 days until participants met criteria for discontinuation of study drug On weeks with Elotuzumab dosing: Tablets, Oral, 28 mg Repeat every 28 days until participants met criteria for discontinuation of study drug Dexamethasone (IV): On weeks without Elotuzumab dosing: Not Applicable (N/A) On weeks with Elotuzumab dosing: Solution, Intravenous (IV), 8 mg, weekly Repeat every 28 days until participants met criteria for discontinuation of study drug Elotuzumab (BMS-901608; HuLuc63): Solution, IV, 10 mg/kg, weekly, on Days 1, 8, 15, 22 (cycles 1&2); Days 1 and 15 (cycles 3 and beyond) Repeat every 28 days until participants met criteria for discontinuation of study drug
- Lenalidomide + Dexamethasone: Lenalidomide: Capsules, Oral, 25 mg, once daily, on Days 1-21 Regimen repeated every 28 days until participants met criteria for discontinuation of study drug Dexamethasone: Tablets, Oral, 40 mg, weekly, on Days 1, 8, 15, 22 Regimen repeated every 28 days until participants met criteria for discontinuation of study drug
Period: Randomized Participants
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Started | 321 | 325
Completed | 319 | 316
Not Completed | 2 | 9
Not completed — Participant no longer meets study criteria | 1 | 1
Not completed — Participant withdrew consent | 1 | 7
Not completed — Adverse event unrelated to study drug | 0 | 1
Period: Treated Participants
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Started (Participants treated) | 318 (1 participant was randomized to treatment E-Ld but received treatment Ld) | 317 (1 participant was randomized to treatment E-Ld but received treatment Ld)
Completed (Participants still on treatment) | 0 | 0
Not Completed | 318 | 317
Not completed — Disease progression | 185 | 185
Not completed — Study drug toxicity | 39 | 45
Not completed — Adverse event unrelated to study drug | 31 | 37
Not completed — Participants request to discontinue study treatment | 28 | 18
Not completed — Administrative reason by sponsor | 13 | 4
Not completed — Other reasons | 14 | 14
Not completed — Participant withdrew consent | 6 | 11
Not completed — Death | 1 | 1
Not completed — Participant no longer meets study criteria | 1 | 1
Not completed — Poor/non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized: all participants randomized to any treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone | Total
Number analyzed (Participants) | 321 | 325 | 646
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.34) | 65.3 (10.26) | 65.7 (9.81)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 134 | 142 | 276
  >= 65 and < 75 years old | 119 | 122 | 241
  >= 75 years old | 68 | 61 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 132 | 261
  Male | 192 | 193 | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 28 | 33 | 61
  Unknown or Not Reported | 288 | 291 | 579
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 264 | 280 | 544
  Black or African American | 13 | 10 | 23
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 31 | 64
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 9 | 4 | 13
  Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Primary definition of Progression-free survival (PFS) defined as the time from randomization to the date of first documented tumor progression or death due to any cause. Participants were censored at the last adequate assessment prior to the start of any subsequent systemic-therapy or at the last adequate assessment prior to 2 missing assessments (> 10 weeks). Participants who died more than 10 weeks after the randomization date and had no on-treatment assessment were censored at the randomization date. Clinical deterioration was not considered progression. The primary analysis of PFS was based on the primary definition using the Independent Review Committee (IRC) tumor assessment using the European Group for Blood and Bone Marrow Transplant (EBMT) criteria. Tumor assessments were made every 4 weeks (±1 week) relative to the first dose of study medication.
Time Frame: From randomization up to 326 events (up to approximately 38 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 321 | 325
Months | 19.35 [16.62 to 22.18] | 14.85 [12.09 to 17.22]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone + Elotuzumab vs Lenalidomide + Dexamethasone; Hazard Ratio of Lenalidomide + Dexamethasone + Elotuzumab to Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.0014, Log Rank; 2-sided p-value for stratified log rank test; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.60 to 0.89]

2. Post Hoc Outcome: Median Progression Free Survival (PFS) - Extended Collection
Description: The time from randomization to the date of first documented tumor progression or death due to any cause. Participants were censored at the last adequate assessment prior to the start of any subsequent systemic-therapy or at the last adequate assessment prior to 2 missing assessments (> 10 weeks). Participants who died more than 10 weeks after the randomization date and had no on-treatment assessment were censored at the randomization date. Clinical deterioration was not considered progression. Tumor assessments were made every 4 weeks (±1 week) relative to the first dose of study medication based on Independent Review Committee (IRC) tumor assessment using the European Group for Blood and Bone Marrow Transplant (EBMT) criteria.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 06-Jul-2018)
Time Frame: From randomization up to to the date of first documented tumor progression or death (up to approximately 85 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 321 | 325
Months | 19.42 [16.62 to 22.31] | 14.92 [12.25 to 17.31]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone + Elotuzumab vs Lenalidomide + Dexamethasone; Hazard Ratio of Lenalidomide + Dexamethasone + Elotuzumab to Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.0005, Log Rank; 2-sided p-value for stratified log rank test; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.60 to 0.87]

3. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) defined as the percentage of participants with a best response on-study of partial response (PR) or better (stringent CR [sCR], complete response [CR], very good partial response [VGPR], and partial response [PR]) based on the Independent Review Committee (IRC) assessment of best response using the European Group for Blood and Bone Marrow Transplant (EBMT) assessment criteria. Participants were censored at the last adequate assessment prior to the start of any subsequent systemic-therapy or at the last adequate assessment prior to 2 missing assessments (> 10 weeks). Participants who died more than 10 weeks after the randomization date and had no on-treatment assessment were censored at the randomization date. Clinical deterioration was not considered progression. Assessments were made every 4 weeks.
Time Frame: From randomization up to approximately 38 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 321 | 325
Percentage of participants | 78.5 [73.6 to 82.9] | 65.5 [60.1 to 70.7]
Statistical Analysis 1: Comparison: Lenalidomide + Dexamethasone + Elotuzumab vs Lenalidomide + Dexamethasone; Ratio of Lenalidomide + Dexamethasone + Elotuzumab to Lenalidomide + Dexamethasone; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by B2 microglobulin (<3.5 mg/L vs >=3.5 mg/L), number of prior lines of therapy (1 vs >=2), and immunomodulatory drug use at randomization; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.36 to 2.78]
Statistical Analysis 2: Comparison: Lenalidomide + Dexamethasone + Elotuzumab vs Lenalidomide + Dexamethasone; Difference of Lenalidomide + Dexamethasone + Elotuzumab minus Lenalidomide + Dexamethasone computed using the method of DerSimonian and Laird (weighted average over the strata); Test type: Superiority; Difference in ORR = 12.7, 95% CI 2-sided [6.2 to 19.3]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death from any cause. If a subject has not died, their survival time will be censored at the date of last contact ("last known alive date"). A subject will be censored at the date of randomization if they were randomized but had no follow-up. (Based on Kaplan Meier estimates)
Time Frame: Randomization to the date of death from any cause (up to approximately 9 years)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 321 | 325
Months | 48.30 [40.34 to 51.94] | 39.62 [33.25 to 45.27]

5. Secondary Outcome: Change From Baseline of Mean Score Pain Severity (BPI-SF)
Description: The change from baseline of the mean score of pain severity at the end of treatment using the Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF is a self administered questionnaire developed to assess the severity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension). The BPI-SF uses 0 ("No pain", "No interference") to 10 ("Pain as bad as you can imagine", "Highest imaginable interference") numeric rating scale.
Time Frame: From baseline up to approximately 38 months
Population: All randomized participants with baseline and end of treatment scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 114 | 152
Score on a scale | 0.52 (2.237) | -0.04 (2.408)

6. Secondary Outcome: Change From Baseline of Mean Score Pain Interference (BPI-SF)
Description: The change from baseline of the mean score of pain interference at the end of treatment using the Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF is a self administered questionnaire developed to assess the severity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension). The BPI-SF uses 0 ("No pain", "No interference") to 10 ("Pain as bad as you can imagine", "Highest imaginable interference") numeric rating scale.
Time Frame: From baseline up to approximately 38 months
Population: All randomized participants with baseline and end of treatment scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
Number analyzed (Participants) | 113 | 150
Score on a scale | 0.95 (2.466) | 0.48 (2.868)

ADVERSE EVENTS:
Time Frame: From first dose up to 60 days post last dose of study therapy (Up to approximately 9 years)
Description: Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed/monitored for the treated population. All-Cause Mortality was assessed for the randomized population.
Arm/Group | Lenalidomide + Dexamethasone + Elotuzumab | Lenalidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 226/321 | 249/325
Serious Adverse Events (participants affected / at risk) | 238/318 | 194/317
Other Adverse Events (participants affected / at risk) | 314/318 | 309/317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Dexamethasone + Elotuzumab (N=318) | Lenalidomide + Dexamethasone (N=317)
Anaemia (Blood and lymphatic system disorders) | 11 | 8
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 4
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 9
Atrioventricular block complete (Cardiac disorders) | 2 | 0
Brugada syndrome (Cardiac disorders) | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 6 | 6
Cataract nuclear (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 12
Diverticulum (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 4 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Disease progression (General disorders) | 15 | 10
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 5 | 4
Hernia (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 25 | 17
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 2
Atypical pneumonia (Infections and infestations) | 3 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 8 | 8
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Catheter site abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 8 | 1
Cerebral aspergillosis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 2
Enteritis infectious (Infections and infestations) | 1 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 4
Genital abscess (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 4 | 1
Herpes zoster reactivation (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 4
Intervertebral discitis (Infections and infestations) | 0 | 1
Large intestine infection (Infections and infestations) | 1 | 0
Listeriosis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 8 | 4
Lung abscess (Infections and infestations) | 0 | 1
Meningitis staphylococcal (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 56 | 40
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 2 | 2
Pneumonia pneumococcal (Infections and infestations) | 3 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 11 | 4
Retinitis (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 8
Septic shock (Infections and infestations) | 2 | 5
Sinusitis (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 5
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 2 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Chemical burn (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 1 | 0
Escherichia test positive (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 1 | 1
Influenza B virus test positive (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Polymerase chain reaction positive (Investigations) | 0 | 1
Viral test positive (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute erythroid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 3
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Dementia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 2
Spinal cord disorder (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Device dislocation (Product Issues) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 11 | 8
Haematuria (Renal and urinary disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Myeloma cast nephropathy (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 5
Renal impairment (Renal and urinary disorders) | 3 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 10 | 4
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 2
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Dexamethasone + Elotuzumab (N=318) | Lenalidomide + Dexamethasone (N=317)
Anaemia (Blood and lymphatic system disorders) | 135 | 118
Leukopenia (Blood and lymphatic system disorders) | 26 | 26
Lymphopenia (Blood and lymphatic system disorders) | 41 | 23
Neutropenia (Blood and lymphatic system disorders) | 114 | 137
Thrombocytopenia (Blood and lymphatic system disorders) | 91 | 72
Cataract (Eye disorders) | 58 | 36
Vision blurred (Eye disorders) | 31 | 18
Abdominal pain (Gastrointestinal disorders) | 44 | 31
Abdominal pain upper (Gastrointestinal disorders) | 30 | 20
Constipation (Gastrointestinal disorders) | 115 | 89
Diarrhoea (Gastrointestinal disorders) | 159 | 122
Dry mouth (Gastrointestinal disorders) | 16 | 10
Dyspepsia (Gastrointestinal disorders) | 36 | 19
Nausea (Gastrointestinal disorders) | 82 | 73
Stomatitis (Gastrointestinal disorders) | 30 | 14
Toothache (Gastrointestinal disorders) | 18 | 11
Vomiting (Gastrointestinal disorders) | 58 | 32
Asthenia (General disorders) | 80 | 54
Chest pain (General disorders) | 28 | 14
Chills (General disorders) | 31 | 12
Fatigue (General disorders) | 154 | 131
Influenza like illness (General disorders) | 27 | 16
Malaise (General disorders) | 19 | 12
Oedema peripheral (General disorders) | 97 | 78
Pain (General disorders) | 17 | 7
Pyrexia (General disorders) | 121 | 74
Bronchitis (Infections and infestations) | 66 | 52
Gastroenteritis (Infections and infestations) | 18 | 9
Herpes zoster (Infections and infestations) | 18 | 5
Influenza (Infections and infestations) | 25 | 17
Lower respiratory tract infection (Infections and infestations) | 32 | 16
Nasopharyngitis (Infections and infestations) | 83 | 60
Oral herpes (Infections and infestations) | 20 | 13
Pharyngitis (Infections and infestations) | 17 | 16
Pneumonia (Infections and infestations) | 30 | 23
Respiratory tract infection (Infections and infestations) | 36 | 32
Rhinitis (Infections and infestations) | 30 | 13
Sinusitis (Infections and infestations) | 23 | 15
Upper respiratory tract infection (Infections and infestations) | 86 | 62
Urinary tract infection (Infections and infestations) | 36 | 31
Viral infection (Infections and infestations) | 18 | 10
Contusion (Injury, poisoning and procedural complications) | 44 | 28
Fall (Injury, poisoning and procedural complications) | 21 | 14
Alanine aminotransferase increased (Investigations) | 25 | 33
Aspartate aminotransferase increased (Investigations) | 21 | 31
Blood creatinine increased (Investigations) | 36 | 27
C-reactive protein increased (Investigations) | 13 | 16
Platelet count decreased (Investigations) | 16 | 5
Weight decreased (Investigations) | 52 | 20
Decreased appetite (Metabolism and nutrition disorders) | 71 | 42
Hyperglycaemia (Metabolism and nutrition disorders) | 61 | 45
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 48 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 67 | 47
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 18 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 19 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 98 | 63
Back pain (Musculoskeletal and connective tissue disorders) | 105 | 97
Bone pain (Musculoskeletal and connective tissue disorders) | 33 | 43
Muscle spasms (Musculoskeletal and connective tissue disorders) | 99 | 85
Muscular weakness (Musculoskeletal and connective tissue disorders) | 42 | 28
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 39 | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 22
Neck pain (Musculoskeletal and connective tissue disorders) | 23 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 64 | 35
Dizziness (Nervous system disorders) | 48 | 38
Headache (Nervous system disorders) | 54 | 29
Hypoaesthesia (Nervous system disorders) | 28 | 12
Neuropathy peripheral (Nervous system disorders) | 51 | 31
Paraesthesia (Nervous system disorders) | 35 | 29
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 39
Taste disorder (Nervous system disorders) | 18 | 14
Tremor (Nervous system disorders) | 30 | 29
Anxiety (Psychiatric disorders) | 26 | 24
Confusional state (Psychiatric disorders) | 18 | 10
Depression (Psychiatric disorders) | 18 | 14
Insomnia (Psychiatric disorders) | 79 | 83
Mood altered (Psychiatric disorders) | 23 | 8
Dysuria (Renal and urinary disorders) | 16 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 109 | 62
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 72 | 60
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 20 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25 | 5
Erythema (Skin and subcutaneous tissue disorders) | 26 | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 38 | 25
Night sweats (Skin and subcutaneous tissue disorders) | 24 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 29
Rash (Skin and subcutaneous tissue disorders) | 63 | 58
Deep vein thrombosis (Vascular disorders) | 19 | 10
Flushing (Vascular disorders) | 16 | 6
Haematoma (Vascular disorders) | 17 | 8
Hypertension (Vascular disorders) | 40 | 23
Hypotension (Vascular disorders) | 33 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.